CLINICAL TRIAL: NCT03197506
Title: Phase II Study of Pembrolizumab (MK-3475) in Combination With Standard Therapy for Newly Diagnosed Glioblastoma
Brief Title: Pembrolizumab and Standard Therapy in Treating Patients With Glioblastoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC1572; NCI-2017-01106 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1572 (Other: Mayo Clinic in Rochester); 16-002965 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2017-06-21; First posted 2017-06-23 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Glioblastoma; Gliosarcoma; Supratentorial Glioblastoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Radiation; pembrolizumab; Radiotherapy; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (pembrolizumab, surgery, temozolomide, radiation) (Experimental): NEOADJUVANT (CYCLE 1): Patients receive pembrolizumab IV over 30 minutes on day 1.
  SURGERY (CYCLE 2): Patients undergo standard of care surgery within days 4-7.
  CONCURRENT (CYCLE 3): Starting 21-35 days after surgery, patients receive pembrolizumab IV over 30 minutes on days 1, 22, and 43 and temozolomide PO daily on days 8-54. Patients also undergo external beam radiation therapy every 5 days per week on days 8-54.
  ADJUVANT (CYCLE 4-8): Within 3-5 weeks after completing radiation therapy, patients receive pembrolizumab IV over 30 minutes on days 1, 22, and 43 and temozolomide PO daily on days 1-5 every 28 days. Treatment repeats every 63 days for up to 5 cycles in the absence of disease progression or unexpected toxicity.
  Interventions: Radiation: External Beam Radiation Therapy; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Radiation: Radiation Therapy; Drug: Temozolomide; Procedure: Therapeutic Conventional Surgery
- Group 2 (pembrolizumab, temozolomide, radiation therapy ) (Experimental): CONCURRENT (CYCLE 1): Starting 21-35 days after surgery, patients receive pembrolizumab IV over 30 minutes on days 1, 22, and 43 and temozolomide PO daily on days 8-54. Patients also undergo external beam radiation therapy every 5 days per week on days 8-54.
  ADJUVANT (CYCLES 2-6): Within 3-5 weeks after completing radiation therapy, patients receive pembrolizumab IV over 30 minutes on days 1, 22, and 43 of cycles 2-5 and 1 and 22 of cycle 6 (up to a total of 17 doses). Patients also receive temozolomide PO daily on days 1-5, 29-33, and 57-61 of cycles 2 and 6, days 22-26 and 50-54 of cycle 3, days 15-19 and 43-47 of cycle 4, days 8-12 and 36-40 of cycle 5. Treatment repeats every 63 days for up to 5 cycles in the absence of disease progression or unexpected toxicity.
  Interventions: Radiation: External Beam Radiation Therapy; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Radiation: Radiation Therapy; Drug: Temozolomide

INTERVENTIONS:
Radiation: External Beam Radiation Therapy — Undergo external beam radiation therapy
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam; Teleradiotherapy; Teletherapy; Teletherapy Radiation
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac; TMZ
Procedure: Therapeutic Conventional Surgery — Undergo surgery
  Arms: Group 1 (pembrolizumab, surgery, temozolomide, radiation)

SUMMARY:
This phase II trial studies the side effects and how well pembrolizumab works in combination with standard therapy in treating patients with glioblastoma. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Drugs used in the chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy beams to kill tumor cells and shrink tumors. Giving pembrolizumab and standard therapy comprising of temozolomide and radiation therapy may kill tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and tolerability of pembrolizumab in combination with standard therapy (surgery, external beam radiation therapy and temozolomide [TMZ] chemotherapy) in patients with newly diagnosed glioblastoma multiforme (GBM). (Neoadjuvant [Group 1]) II. To assess the 18 month overall survival rate of pembrolizumab in combination with standard therapy (surgery, external beam radiation therapy and TMZ chemotherapy) in patients with newly diagnosed glioblastoma multiforme (GBM). (Adjuvant [Group 2])

SECONDARY OBJECTIVES:

I. To assess adverse events (AE) and toxicity profile of pembrolizumab in combination with standard therapy in patients with newly diagnosed GBM.

II. To assess time to progression in patients treated with pembrolizumab in combination with standard therapy in patients with newly diagnosed GBM. (Adjuvant only) III. To assess progression-free survival in patients treated with pembrolizumab in combination with standard therapy in patients with newly diagnosed GBM. (Adjuvant only) IV. To assess time to treatment failure in patients treated with pembrolizumab in combination with standard therapy in patients with newly diagnosed GBM. (Adjuvant only)

CORRELATIVE RESEARCH OBJECTIVES:

I. To assess the tumor PD-1/PD-L1 expression and inflammatory microenvironment profile by comparing PD-1/PD-L1 expression and T lymphocyte/monocytic infiltrates before and after administration of pembrolizumab treatment. (Neoadjuvant only) II. To assess the peripheral immunophenotype profile and GBM-associated antigen-specific T cell responses before and after receiving pembrolizumab treatment in combination with standard therapy.

OUTLINE: Patients are assigned to 1 of 2 groups.

GROUP 1:

NEOADJUVANT (CYCLE 1): Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1.

SURGERY (CYCLE 2): Patients undergo standard of care surgery within days 4-7.

CONCURRENT (CYCLE 3): Starting 21-35 days after surgery, patients receive pembrolizumab IV over 30 minutes on days 1, 22, and 43 and temozolomide orally (PO) daily on days 8-54. Patients also undergo external beam radiation therapy every 5 days per week on days 8-54.

ADJUVANT (CYCLE 4-8): Within 3-5 weeks after completing radiation therapy, patients receive pembrolizumab IV over 30 minutes on days 1, 22, and 43 and temozolomide PO daily on days 1-5 every 28 days. Treatment repeats every 63 days for up to 5 cycles in the absence of disease progression or unexpected toxicity.

GROUP 2:

CONCURRENT (CYCLE 1): Starting 21-35 days after surgery, patients receive pembrolizumab IV over 30 minutes on days 1, 22, and 43 and temozolomide PO daily on days 8-54. Patients also undergo external beam radiation therapy every 5 days per week on days 8-54.

ADJUVANT (CYCLES 2-6): Within 3-5 weeks after completing radiation therapy, patients receive pembrolizumab IV over 30 minutes on days 1, 22, and 43 of cycles 2-5 and 1 and 22 of cycle 6 (up to a total of 17 doses). Patients also receive temozolomide PO daily on days 1-5, 29-33, and 57-61 of cycles 2 and 6, days 22-26 and 50-54 of cycle 3, days 15-19 and 43-47 of cycle 4, days 8-12 and 36-40 of cycle 5. Treatment repeats every 63 days for up to 5 cycles in the absence of disease progression or unexpected toxicity.

After completion of study treatment, patients are followed up at 30 days, every 3 months until progressive disease, then every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Histological confirmation of supratentorial glioblastoma (also known as astrocytoma grade IV, gliosarcoma)

  * NOTE: Grade IV IDH-mutant astrocytoma is also allowed
* Neoadjuvant patients only: Have an enhancing mass on magnetic resonance imaging (MRI) amenable to > 90% resection of contrast-enhancing tumor (as determined by the neurosurgeon pre-operatively) and histological diagnosis of glioblastoma or astrocytoma from a prior biopsy or surgery

  * NOTE: Biopsy or subtotal resection must have been =< 43 days prior to registration
* Neoadjuvant patients only: Willing to undergo craniotomy and resection of their brain tumor at Mayo Clinic in Rochester, Minnesota (MN)
* Adjuvant patients only: Must have undergone craniotomy and resection of their brain tumor =< 6 weeks prior to registration
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
* Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 28 days prior to registration)
* Platelet count >= 100,000/mm^3 (obtained =< 28 days prior to registration)
* Hemoglobin >= 9.0 g/dL without transfusion or erythropoietin (EPO) dependency (=< 7 days prior to assessment) (obtained =< 28 days prior to registration)
* Prothrombin time (PT) =< 1.5 x upper limit of normal (ULN) unless patient is receiving anticoagulant therapy and PT or partial prothrombin time (PTT) is within therapeutic range of intended use of coagulants (obtained =< 28 days prior to registration)
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless patient is receiving anticoagulant therapy and PT or PTT is within therapeutic range of intended use of coagulants (obtained =< 28 days prior to registration)
* Albumin >= 2.5 mg/dL (obtained =< 28 days prior to registration)
* Total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for patients with total bilirubin levels > 1.5 x ULN (obtained =< 28 days prior to registration)
* Aspartate transaminase (AST) AND alanine transaminase (ALT) =< 2.5 x ULN (obtained =< 28 days prior to registration)
* Creatinine =< 1.0 x ULN OR measured or calculated creatinine clearance (per institutional standard) must be >= 60 ml/min (obtained =< 28 days prior to registration)
* Negative pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only (POCBP)

  * NOTE: Serum or urine pregnancy test allowed; if urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* POCBP must be willing to use adequate contraception starting with first dose through 120 days after last dose
* Provide written informed consent
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)

  * Note: During the active monitoring phase of a study (i.e., active treatment and observation), participants must be willing to return to the consenting institution for follow-up
* Willing to provide tissue and blood samples for correlative research purposes

Exclusion Criteria:

* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ adequate contraception
* Neoadjuvant patients only: Signs or symptoms of life-threatening raised intracranial pressure: as defined by the treating neurosurgeon, including severe headache, nausea, decreasing level of consciousness, precluding 4-7 day delay in scheduling neurosurgery
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy =< 5 years prior to registration

  * EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix
  * NOTE: If there is a history or prior malignancy, the patient must not be receiving other specific treatment for their cancer
* History of myocardial infarction =< 6 months prior to registration, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs; NOTE: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Known history of active TB (Bacillus tuberculosis)
* Received a live vaccine =< 30 days prior to registration
* History of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Hypersensitivity to pembrolizumab or any of its excipients
* Received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* Received or planning to receive Optune device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2028-06-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLT) (Group 1) | Up to 189 days (3 cycles of treatment)
  A DLT will be defined as an adverse event attributed (definitely, probably, or possibly) to pembrolizumab per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Overall survival (OS) (Group 2) | 18 months
  Defined as the time from beginning study therapy to death due to any cause. Will be assessed by the number of patients who are alive up to 18 months after beginning study therapy.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 5 years
  The number and severity of all adverse events will be tabulated and summarized in this patient population. Specifically, the overall toxicity percentages for Grade 3 or higher adverse events considered at least possibly related to treatment will be calculated and reported. All other adverse event analysis will be exploratory and hypothesis generating.
Time until any treatment related adverse event | Up to 5 years
  Will be summarized descriptively.
Time until treatment related grade 3+ adverse event | Up to 5 years
  Will be summarized descriptively.
Time until hematologic nadirs | Up to 5 years
  Will assess the time until hematologic nadirs (white blood cell count, absolute neutrophil count, platelets) and will be summarized descriptively.
Time to progression (Group 2) | Up to 5 years
  Defined as the time from start of study treatment to disease progression. Will be assessed using the immunotherapy response assessment for neuro-oncology (iRANO) criteria.
Progression-free survival (Group 2) | Up to 5 years
  Defined as the time from starting study treatment to the date of disease progression or death resulting from any cause, whichever comes first. Will be assessed according to iRANO criteria.
Time to treatment failure (Group 2) | Up to 5 years
  Defined as the time from beginning study therapy to documentation of disease progression, unacceptable adverse event(s), or refusal to continue participation by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Ian F. Parney, MD, PhD, Principal Investigator — Mayo Clinic in Rochester
Locations (3):
- United States (3):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials